CLINICAL TRIAL: NCT05759975
Title: Effectiveness of Extraoral Photobiomodulation Protocols in Management of Oral Adverse Effects in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Effectiveness of Extraoral Photobiomodulation in Management of Oral Adverse Effects in Patients Undergoing HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Manoela Domingues Martins, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBM and MO HSCT
Record Dates: First submitted 2022-12-30; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Oral Mucositis; Hematopoietic Neoplasm; Xerostomia; Hyposalivation
MeSH Terms: conditions — Stomatitis; Hematologic Neoplasms; Xerostomia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two groups for the duration of the study. Group I (PBMI, n=21) photobiomodulation intraoral with a low potency laser, and Group II: photobiomodulation with high power extraoral unfocused laser with 1 W power (PBME, n=21).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know the laser protocol of each patient (single blind) .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraoral photobiomodulation (PBMI) (Active Comparator): The protocol will be performed daily by a single trained professional from the first day of conditioning until D + 5 after bone marrow transplantation or while lesions are present.
  PBMI protocol will use the indium-gallium-aluminium-phosphorus diode laser (InGaAlP) (DUO® - MMOptics Ltda, São Carlos, Brazil). Four anatomical areas will be irradiated perpendicularly in the buccal mucosa through several anatomical points with a distance of approximately 1 cm between them, in order to cover the largest area per cm² by region.
  Application points:
  * Buccal mucosa: 9 points each side: bite line on cheeks and upper and lower internal buccal vestibule (18 points).
  * Tongue: 4 points on each side, on the lateral and ventral edge (8 points).
  * Floor of the mouth: 1 point on each side (2 points)
  * Upper and lower lips: upper and lower lips (lip redness), bottom of upper and lower sulcus and buccal commissure, right and left sides (4 points).
  * Soft palate: right and left side (2 points)
  Interventions: Device: Photobiomodulation therapy (intraoral)
- Extraoral photobiomodulation (PBME) (Active Comparator): The protocol will be performed daily by a single trained professional from the first day of conditioning until D + 5 after bone marrow transplantation or while lesions are present.
  A gallium-aluminum arsenide diode laser (Gemini® manufactured by Azena Medical, LLC, distributed by Ultradent Products, Inc.) with double wavelength 810 + 980 nm, previously standardized and calibrated for extraoral application by the measurement of potency (Coherent Inc, Santa Clara, CA). The equipment will be programmed with 1 W of power. The application points will be carried out perpendicularly on the face.
  Application points:
  * 4 points on each cheek (2 on the right and 2 on the left)
  * 1 on lips; patients with sealed lips being possible to cover the upper and lower lip
  * 5 points in the cervical region (2 in the right submandibular space and 2 in the left submandibular space and submental space in the midline).
  Interventions: Device: Photobiomodulation therapy (extraoral)

INTERVENTIONS:
Device: Photobiomodulation therapy (intraoral) — Intraoral photobiomodulation therapy (660nm, 100mW, 10 J/cm 2 , 3 s/point) for the management of oral side effects related during hematopoietic stem cell transplantation (HSCT). Mainly in the decrease of oral OM rates and OM severity, healing of OM ulcers and pain relief. Second, evaluate quality of life,hyposalivation/xerostomia, functional evaluation and dysfagia, in the arm. All results obtained in the group will be compared with the other arm.
  Arms: Intraoral photobiomodulation (PBMI)
Device: Photobiomodulation therapy (extraoral) — Extraoral photobiomodulation therapy (810 + 980 nm, 1 W, 6.11 J/cm2 , 30 s/point) for the management of oral side effects related during hematopoietic stem cell transplantation (HSCT). Mainly in the decrease of oral OM rates and OM severity, healing of OM ulcers and pain relief. Second, evaluate quality of life,hyposalivation/xerostomia, functional evaluation and dysfagia, in the arm. All results obtained in the group will be compared with the other arm.
  Arms: Extraoral photobiomodulation (PBME)

SUMMARY:
Patients undergoing hematopoietic cell transplantation (HSCT) receive high doses of chemotherapy with or without radiotherapy to eradicate the underlying disease, which induces a series of adverse effects, including in the oral cavity. Among the most common oral lesions is oral mucositis (OM), which has been associated with greater morbidity and important biological and economic impact.Currently, photobiomodulation (PBM) with intraoral application has been recommended for the prevention of OM, however, few studies have evaluated the impact of its extraoral use.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effectiveness of extraoral PBM using unfocused high-power laser compared to intraoral PBM with low-power laser in the management of OM, mouth pain, functional capacity, development and duration of hyposalivation and xerostomia and quality of life. This is a multicenter, randomized, single blind clinical trial to be conducted at the Hospital de Clínicas de Porto Alegre (HCPA) and at the AC Camargo Cancer Center Hospital.

All patients who accept participate of the study will assign an informed consent form. For data management, the REDcap® software will be used, where all forms referring to patients evaluation will be incorporated. 42 patients will be selected who will undergo HSCT regardless of the underlying disease. Subsequently, upon accepting participation in the study, participants will undergo a sequential allocation using the R shiny summary statistics ® software by the variables of gender, age, type of HSCT and type of conditioning and will be allocated into 2 groups: Group I : intraoral photobiomodulation (660nm, 100mW, 10 J/cm 2 , 3 s/point) (PBMI, n=21) and Group II: extraoral photobiomodulation (810 + 980 nm,1 W,6.11 J/cm 2, 30 s/point) with high power extraoral unfocused laser with 1 W power (PBME, n=21). In both arms, the patients will receive photobiomodulation therapy from the the beginning of the conditioning until D + 5 after HSCT procedure. If any patient presenting or developing lesion after D + 5, this patient will receive the photobiomodulation protocol stipulated in your respective group util occur the healing of the lesion.

The study will be carried out by a dental surgeon who will carry out the initial assessment and reassessments (blinded to the groups) and another who will carry out the application of the PBM. Patients will be evaluated daily from the beginning of the conditioning until the bone marrow grafting or while there are oral lesions.

If they do not develop lesions, after bone marrow grafting, the patients will be evaluated weekly until hospital discharge. After clinical exam, grade and OM severity will be evaluated, after that, classified according WHO and NCI scale, pain assessment (VAS and NRS-101) and functional assessment, until D + 5 after HSTC procedure. The evaluation of xerostomia/hyposalivation (stimulated and non-stimulated salivary flow and xerostomia inventory) and quality of life will be performed in three moments, at the beginning of the conditioning, on the day of the HSCT and on the bone marrow marrow grafting day.

Saliva samples will be collected with SWABS, to futures microbioma analysis. The statistical analyzes will be carried out in the PASW 18.0 program, initially the evaluation of the data distribution will be carried out from the application of the Shapiro-Wilk and Kolmogorov-Smirnov tests.

If from the application of these tests, the data show normal distribution (p>0.05), the t test will be used. If the distribution proves to be non-normal from the application of the test (p<0.05), the Wilcoxon test will be used. The p-value will be set to 5%. Logistic regression will be used in fitted models to estimate the probability of occurrence of OM (dependent variable) in relation to clinical demographic variables (independent variables).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and scheduled for autologous or allogeneic HSCT.
* Patients undergoing myeloablative conditioning regimen

Exclusion Criteria:

* Patients previously submitted to autologous or allogeneic HSCT
* Patients on a non-myeloablative conditioning regimen
* Patients on a reduced-intensity conditioning regimen

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis evaluation according WHO scale | 16 months
  The measurement of mucositis will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
  Mucositis will be scored according to WHO criteria: grade 0 (none), grade I (oral soreness, erythema), grade II (oral erythema, ulcers, solid and liquid diet tolerated), grade III (oral ulcers, liquid diet only), and grade IV (oral diet impossible).
Oral Mucositis evaluation according NCI scale | 16 months
  The measurement of mucositis will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
  The National Cancer Institute (NCI) scale (NCI - Common Terminology Criteria for Adverse Events) will be performed: grade I (mucosal erythema), grade II ( patchy ulcerations with pseudomembranes), grade III (confluent ulceration or pseudomembranes, bleeding with minor trauma), and grade IV (tissue necrosis, significant spontaneous bleeding)

SECONDARY OUTCOMES:
Pain evaluation (VAS) | 16 months
  Evaluation of pain, will be employed the visual analogical scale (VAS). Pain evaluation will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
  VAS scale will be represented by a 10 centimeters line, 0 corresponding no pain ranging up to 10 worst pain possible. The patient will be instructed to slide the marker though 10 centimeters line.
Pain evaluation (NRS-101) | 16 months
  Also, Numeric Rating Scale (NRS-101) will be employed. Pain evaluation will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
  NRS-101, the patients will be instructed to assign one number between 0 (no pain) varying until 100 (worst pain possible).
Functional evaluation | 16 months
  Analysis of chewing, swallowing, liquid intake and taste alteration. Responses will be scored daily ranging from 0 - no difficulty, to 4 - impossible to accomplish. The functional evaluation will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
Dysfagia | 16 months
  Will be taken into account - total absence of dysphagia, dysphagia to solid food and dysphagia to any liquid or solid food. Dysfagia evaluation will be performed daily from the beginning of the conditioning therapy until the bone marrow grafting or while there are oral lesions.
Hyposalivation/xerostomia | 16 months
  * Non-stimulated saliva: the patient will be instructed to sit down calmly, tilt the head down, a millimeter collection tube, positioned below the lower lip, for 5 minutes, all the saliva produced will be deposited in the tube
  * Stimulated saliva: the patient will remain seated, with the head tilted forward and the collection of non-stimulated saliva will be performed immediately afterwards. With the patient in the same position, he will chew a silicone sialogogue provided and all the saliva produced during the 5-minute period will be dispensed into another tube identical to the first one. The measurement of the volume of saliva collected will be considering the graduation of the tube.
  Parameters: < 0.1 ml/min will be considered hyposalivation for unstimulated, < 0.7 ml/min for stimulated salivation
  Saliva samples will be collected at the beginning of the conditioning, on the day of the HSCT and on the bone marrow marrow grafting day.
Evaluation of the the quality of life | 16 months
  The Oral Health Impacts Profile questionnaire (OHIP -14) will be employed. Quality of life will be evaluated at the beginning of the conditioning, on the day of the HSCT and on the bone marrow marrow grafting day.
  OHIP is a questionnaire that measures people's perception of the social impact of oral disorders on their well-being. Fourteen items of OHIP are divided into seven dimensions; functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability and handicaps.
  The responses are rated on a 5-point Likert scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = fairly often; 4 = very often/every day. The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better quality of life.
Measure Time | 16 months
  The measure of the time application will be take with a timer during all photobiomodulation sessions
Evaluation of oral health | 16 months
  To assess the impact of treatment on oral health, the manual of epidemiological studies for oral health surveys proposed by the World Health Organization (WHO) will be used. The community periodontal index (CPI) will be used, evaluating two indicators of periodontal condition: gingival bleeding and periodontal pockets (adopting index teeth to record attachment loss).
  An evaluation of the dental condition will also be carried out.
  Oral health will be evaluated at the beginning of the conditioning, on the day of the HSCT, on the bone marrow marrow grafting day, one year and two years after bone marrow grafting.
Saliva analysis | 16 months
  Saliva samples will be collected through SWAB friction in buccal mucosa. After that, the SWABS will be emerged in a buffering saline solution. The tubes will be centrifuged for five minutes at 5000 rpm and the precipitates will be collected. Samples will be frozen in liquid nitrogen and immediately stored at -80 °C until the DNA extraction step.

CONTACTS AND LOCATIONS:
Overall Officials: Manoela D Martins, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Fábio A Alves, PhD, Study Chair — A.C. Camargo Cancer Center
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the outcomes, for one year.
Access Criteria: If formally solicited and referenced by the researcher interested